CLINICAL TRIAL: NCT03398603
Title: Is the Concentration of Anti-Muellerian Hormon (AMH) Depending on the Menstrual Cycle?
Acronym: Bicycle
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Roche Diagnostic Ltd. (Industry)
Responsible Party: Principal Investigator, Christian De Geyter, Professor, University Hospital, Basel, Switzerland
Other Study IDs: 2016-01824
Record Dates: First submitted 2017-12-26; First posted 2018-01-12 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Ovarian Failure
Keywords: AMH measurement "ElecSys"
MeSH Terms: interventions — Blood Specimen Collection; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — For screening titer of hepatitis B/C- and HIV is measured once
  On every second day of two non-consecutive menstrual cycles we take encoded blood samples and measure the AMH value with the "ElecSys" method as well as the hormons LH, FSH, Estradiol und Progesterone
  On every second day of two non-consecutive menstrual cycles we take an encoded vaginal 3D ultrasound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 25 women with age of 18-25 years
  Interventions: Procedure: blood sample and ultrasound
- Group 2: 25 women with age of 26-40 years
  Interventions: Procedure: blood sample and ultrasound

INTERVENTIONS:
Procedure: blood sample and ultrasound — When included in the study blood samples and ultrasound are taken every second day of the first and third menstrual cycle after inclusion.

SUMMARY:
The developement of a new, stable measurement of the Antimuellerian Hormon (AMH) together with Roche Diagnostics International (Rotkreuz, CH) shall enable an automized and timely measurement of AMH values in blood samples.

DETAILED DESCRIPTION:
An important requirement for the use of the new measurement to determine the AMH concentration is the stability of the AMH level over the menstrual cycle. So far the unbiased AMH concentration is the most important argument to manage this parameter.

There are several studies, which give different professional opinions of the AMH concentration depending on the phase of the menstrual cycle. Some authors came to the conclusion that the AMH concentration over the menstrual cycle is constant, others described significant fluctuations. It is unclear, if the described fluctuation is relevant for the interpretation of the ovarian reserve. Recently it could be shown, that intraindividual fluctuations of joung women during the menstrual cycle is stronger, which means that the measurement of AMH in this age is less secure.

The primary goal of the study is to evaluate, if the new AMH measurement with the ElecSys method delivers stable values over the menstrual cycle.

The secondary goal of the study is to determine whether there are any fluctuations in the number of antral follicles as given by 3D ultrasound.

For this reason we are recruiting a group of 50 women within two categories of age to measure eventually changes in AMH- concentration during their menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Regular natural menstrual cycle between 24 and 32 days
* Body Mass Index (BMI) between 19 and 26 kg/m2
* Negative serum titer for HIV, Hepatitis B and Hepatitis C
* Non-smoker
* Willingness to visit the clinic every second day of two non-consecutive menstrual cycles.

Exclusion Criteria:

* Intake of hormonal medication like contraceptives
* Pregnancy/breast feeding
* Known infertility
* Known former or actual hormonal disorder
* Polycystic ovarial syndrom (PCOS)
* Participation on another clinical trial during the last 3 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 healthy female probands
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-10-13 (Actual)

PRIMARY OUTCOMES:
between cycle reliability of ovarian reserve assessment based on AMH serum concentration | 3 months
  stabile assessment of ovarian reserve with AMH (pmol/l) in blood

SECONDARY OUTCOMES:
number of ovarian follicles as made visible by 3D ultrasound | 3 months
  Fluctuations of antral follicle count during different menstrual cycles

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Geyter, Prof., Principal Investigator — USB
Locations (1):
- Klinik für Gyn. Endokrinologie und Reproduktionsmedizin der Frauenklinik des Universitätsspitals, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biniasch M, Laubender RP, Hund M, Buck K, De Geyter C. Intra- and inter-cycle variability of anti-Mullerian hormone (AMH) levels in healthy women during non-consecutive menstrual cycles: the BICYCLE study. Clin Chem Lab Med. 2021 Oct 29;60(4):597-605. doi: 10.1515/cclm-2021-0698. Print 2022 Mar 28. PMID 34717057